CLINICAL TRIAL: NCT06272916
Title: Comparison of the Effect of Aminophylline, Magnesium Sulphate and Placebo in Prevention of Post Dural Puncture Headache in Parturient Undergoing Caesarean Section. A Double-blind Placebo Controlled Trial.
Brief Title: Comparison of the Effect of Aminophylline, Magnesium Sulphate and Placebo in Prevention of Post Dural Puncture Headache in Parturient Undergoing Caesarean Section.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Mohamed Abdelbary Ebrahim, doctor, Assiut University
Other Study IDs: Effect drugs on headache inCS
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Aminophylline; Magnesium Sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sample size of 630 cases was calculated, divided equally into three groups.: For sample size calculation using Yousefshahi et al. (14) as a reference, a sample size of 630 cases was calculated, divided equally into three groups. This sample size achieves 80% power when the effect size is moderate (=0.12) and using 2 degrees of freedom Chi-Squared test with a significant level of 0.05. Using computer generated randomization program, patients were randomly divided into three equal groups.
  Group 1: patient received 100 ml IV infusion of normal saline (control group). Group 2: patient received Aminophylline 1.5 mg/kg IV infusion diluted in normal saline with a total volume of 100 ml.
  Group 3: patient received 50 mg/ kg Magnesium sulfate IV infusion diluted in normal saline with a total volume of 100ml.
  Interventions: Drug: Aminophylline , magnesium sulphate and placebo

INTERVENTIONS:
Drug: Aminophylline , magnesium sulphate and placebo — Comparison of the Effect of Aminophylline, Magnesium Sulphate and Placebo in Prevention of Post Dural Puncture Headache in Parturient Undergoing Caesarean Section

SUMMARY:
This study will be conducted to better comprehend the effect of aminophylline in comparison to magnesium sulphate on preventing and/or treating PDPH.

DETAILED DESCRIPTION:
Delivery by cesarean section (CS) is becoming more frequent and is one of the most common operative procedures performed worldwide. In the USA a CS rate of 26% for all births is reported (1). According to the data by the Central Agency for Public Mobilisation and Statistics (CAPMAS) on the Health of the Egyptian Family (HEF) in late August, C-section births increased to 72 percent in 2021. (2) The postpartum period is marked by the presence of post- dural puncture headache (PDPH) which is an unpleasant emotional and sensory experience. Therefore, any form of intervention that leads to improvement in pain/headache relief can positively impact on patients satisfaction and prevent long hospital stay.

Spinal anesthesia remains the most common analgesic and anesthetic modality in women undergoing CS. It has a worldwide acceptance; it is very reliable and safe as a form of obstetrics anesthesia. Spinal anesthesia also has a fast onset of action and its use is efficacious (3). Although, spinal anesthesia has a generally acceptable complication rate, PDPH has remained its major drawback and unpleasant complication. This complication is especially noticeable few hours after the procedure (4). Although there is no clear pathophysiologic mechanism for PDPH, many treatment options used frequently in clinical practice to prevent or treat headache have been tried but currently there is still no approach that has been shown to offer complete prevention or treatment of the PDPH. Apart from the choice of insertion technique, optimal needle size and tip (5).

The incidence of PDPH has been estimated between 1% and 40% based on the gauge and orientation of needles, the operator proficiency, etc. The incidence rate of PDPH can also be associated with the type of lumbar puncture.(6) Despite that the therapeutic mechanism of aminophylline on PDPH is not fully described yet (7), some studies suggest that it might be responsible for blocking adenosine receptors, constricting blood vessels, and blocking pain transmission. It also seems that aminophylline can increase the intracellular levels of cyclic adenosine monophosphate. Furthermore, calcium uptake by the endoplasmic reticulum of endothelial cells might be suppressed with the administration of aminophylline; this process induces CSF secretion.

Although the precise mechanism is uncertain, magnesium sulfate's ability to function as a noncompetitive antagonist of (NMDA) receptors among peripheral tissues as well as the central nervous system explains the analgesic effects. It also affects how much intracellular calcium is present (8).

ELIGIBILITY:
Inclusion Criteria:

* All parturient who underwent cesarean section under spinal anesthesia.
* Patients who are willing to participate in the trial gave an informed consent.
* ASA physical status II.
* The age ranged from 20 to 40.
* Body Mass Index (BMI) ranged from 25 to 30 kg/m2.

Exclusion Criteria:

* Patient refusal.
* Allergy to the studied drugs.
* Patients with contraindications to spinal anesthesia.
* Those with past history of chronic headache or recent onset of acute headache were excluded.
* Women who had multiple punctures (>2) during the spinal anesthesia procedure were excluded from the study.
* Patients with advanced decompensated cardiac, renal, hepatic disease.

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: All parturient who underwent cesarean section under spinal anesthesia.
  * Patients who are willing to participate in the trial gave an informed consent.
  * ASA physical status II.
  * The age ranged from 20 to 40.
  * Body Mass Index (BMI) ranged from 25 to 30 kg/m2.
Sampling Method: Non-Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Effect of the study drugs on the incidence and severity of PDPH | 100ml of the prepared study drug intravenously immediately after the baby was delivered and umbilical cord was clamped.